CLINICAL TRIAL: NCT04102046
Title: Assesment of Quality of Life by Functional Independance Score in Hemophilia Patients
Brief Title: Quality of Life in Hemophilia by Clinical Scoring System (FISH)Score
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shymaa Saber, Assiut manqabad, Assiut University
Other Study IDs: FISH score in hemophilia
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2019-09

CONDITIONS: Hemophilia Arthropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To asses quality of life in patients with hemophilia clinically.-

-To avoid or minimize structural damage to goints and muscles by making patients aware of importance of rehabilitation

DETAILED DESCRIPTION:
Hemophilia is a blood-clotting disorder caused by a deficiency in factor VIII (FVIII) or factor IX (FIX), which manifests itself through bleeding in the muscles and joints [1].

There are three categories, depending on the percentage of the blood-clotting factor: severe hemophilia (<1% FVIII/IX), characterised by spontaneous bleeding; moderate hemophilia (1-5% FVIII/FIX), with bleeding from slight injuries; and mild hemophilia (>5-40% FVIII/FIX) with bleeding during surgical procedures or from severe injuries(2).(3) Hemophilia C (a deficiency of Factor XI) is encountered, but its effect on clotting is far less pronounced than A or B Hemophilic arthropathy of the ankle causes pain and deterioration in gait, causing disability. Although some physiotherapy modalities are effective in the management of acute bleeding, the results are unknown in chronic arthropathy Due to the progression of hemophilic arthropathy and the resulting deterioration of the joint, deformities such as the estriction of motion (4). Physiotherapy through the RICE method (Rest, Ice, Compression, and Elevation) has been described for the improvement of acute joint injuries (5)as well as in the management of hemarthrosis in patients with hemophilia (6) Treatment of the ankle with physical therapy is complicated because it involves a small joint surface that bears significant ranges of body weight and the joint limitation alters biomechanical movement during walking(7) Prevention of musculoskeletal morbidity is an important objective in the treatment of hemophilia. Efficacy of such therapy has classically been measured by quantifying the extent of arthropathy using a joint scoring (8)(9)

Design of the Functional Independence Score in Hemophilia

Patients with hemophilia and their therapists were asked to list activities that could be affected by hemophilia. These were categorized according to the International Classification of Functioning, Disability and Health (ICF) (10)Activities that were considered unsafe to perform were excluded from the assessment. Other activities such as the use of transport, education and employment - that could not be assessed objectively in the clinic were also excluded. We finally included seven activities under three categories - self-care, transfers and locomotion (Table 1). Each activity was graded from 1 to 4 according to the amount of assistance required to perform the activity. Each activity and level of independence was clearly defined to reduce interobserver variation.core from 1 to 4 in each area:

1. = the subject is unable to perform the activity, or needs complete assistance to perform the activity;
2. = the subject needs partial assistance/aids/modified (9) (10) instruments/modified environment to perform the activity;
3. = the subject is able to perform the activity without aids or assistance, but with slight discomfort. He is unable to perform the activity like his healthy peers 11 4= the subject is able to perform the activity without any difficulty like other healthy pears

ELIGIBILITY:
Inclusion Criteria:

* congenital Hemophilia A and B patients more than 18 years old

Exclusion Criteria:

* All hemophilia patient less than 18 years old
* Patients with other bleeding disorders
* Patients with other comorbidities that can affect joint function as collagen disease
* Patients on steroids or non-steroidal analgesics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemophilia A and B with goint affection
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-06-28 (Estimated); Primary Completion 2020-09-22 (Estimated); Study Completion 2020-10-10 (Estimated)

PRIMARY OUTCOMES:
Quality of life in hemophilia | One year
  Assesment of quality of life by functional independance score in hemophilia

CONTACTS AND LOCATIONS:
Overall Officials: Osama A Ibrahim, professor, Principal Investigator — Unafifiliated

REFERENCES:
- [Background] Cuesta-Barriuso R, Gomez-Conesa A, Lopez-Pina JA. Physiotherapy treatment in patients with hemophilia and chronic ankle arthropathy: a systematic review. Rehabil Res Pract. 2013;2013:305249. doi: 10.1155/2013/305249. Epub 2013 Aug 12. PMID 23997955
- [Background] Poonnoose PM, Manigandan C, Thomas R, Shyamkumar NK, Kavitha ML, Bhattacharji S, Srivastava A. Functional Independence Score in Haemophilia: a new performance-based instrument to measure disability. Haemophilia. 2005 Nov;11(6):598-602. doi: 10.1111/j.1365-2516.2005.01142.x. PMID 16236109